CLINICAL TRIAL: NCT01195857
Title: Assessment of Subject Use of the Rebiject II Injection Device According to Nurse Examination of Subject Accuracy in 10 Steps as a Dummy Demonstration
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR701068-512
Record Dates: First submitted 2010-08-31; First posted 2010-09-06 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rebif; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating disease of the central nervous system (CNS) and is one of the most common causes of neurological disability in young adults. Rebif is licensed in the United Kingdom for the treatment of relapsing MS and is given 3 times per week by subcutaneous injection. The Rebiject II device is an autoinjector which allows patients easier administration of their Rebif injections.

Prior to treatment, patients receive training on the use of the device and its maintenance. Currently, all treatments for MS are injectable and require long term patient commitment. Rebiject has been developed to improve patient convenience and comfort but does require multiple steps to be carried out in order for the injection to be delivered correctly. Reports from our local call centre and nurse advisors suggest that inaccuracies of use with the Rebiject device are common. By raising awareness of the level of inaccuracy and determining which steps patients are most likely not to complete correctly, modified training programs or modifications to current subject training may be put into place to address these issues. It is also important to demonstrate the link between poor use of the medication device and increased relapse rates or increased injection site reactions.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsing remitting multiple sclerosis and currently receiving Rebif treatment and using the Rebiject II injection device
* Be under regular review by a MS nurse
* Be aged 18 or above
* Be willing and able to participate in the trial and to have provided written informed consent

Exclusion Criteria:

* Receiving disease modifying therapy other than Rebif
* Receiving Rebif but not using the Rebiject II injection device
* Do not self inject
* Are unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing remitting multiple sclerosis who are currently receiving Rebif treatment and using the Rebiject II injection device who are under regular review by a Multiple Sclerosis nurse.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who correctly use the Rebiject II injection device based on reaching all correct injection steps as assessed by a nurse | up to 6 month

SECONDARY OUTCOMES:
Most common 3 steps for error with the Rebiject II injection device out of the ten step checklist | up to 6 month
Correlation with recent training within the last 6 months | up to 6 month
Correlation with disease control (relapse rate) | up to 6 month
Length of time on treatment | up to 6 month
Presence of injection site reactions | up to 6 month
Cognitive impairment | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gillian L Shepherd, MD, MRCP, Study Director — Merck Serono Limited, UK

REFERENCES:
- [Result] Caroline D'Arcy, Laura Parkes, Gillian Shepherd British Journal of Neuroscience Nursing, Vol. 8, Iss. 1, 26 Feb 2012, pp 25 - 31